CLINICAL TRIAL: NCT05763758
Title: Spatiotemporal Thalamocortical Alterations Underlie Experimental and Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Florida State University (Other)
Responsible Party: Principal Investigator, Jian Kong, Principal investigator, Massachusetts General Hospital
Other Study IDs: 2022p003171
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Experimental Pain; Low Back Pain
Keywords: EEG, fMRI, thalamus, pain, experimental pain, low back pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy participants will undergo multimodal neuroimaging during resting state, no-pain and painful tonic pressure presentation. At FSU, EEG and fMRI will be simultaneously acquired. At MGH, sequential MRI and MEG/EEG will be acquired.
  Interventions: Other: No intervention
- Patients with chronic low back pain: Subjects with chronic low back pain (cLBP) patients will undergo multimodal neuroimaging during resting state, no-pain and painful tonic pressure presentation. The study will only be performed at MGH, sequential MRI and MEG/EEG will be acquired.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention involved in this study

SUMMARY:
This study aims to identify spatiotemporal alterations in thalamocortical circuitry functioning in both healthy subjects and patients with chronic pain, combining multimodal neuroimaging.

DETAILED DESCRIPTION:
Investigators will pursue this goal in both experimental and clinical models at two sites (Florida State U/FSU & Mass General Hospital/MGH), implementing parallel enrollment of large and diverse samples (140 healthy participants and 60 patients with chronic low back pain/cLBP). Leveraging the fully developed multimodal neuroimaging methodology-simultaneous EEG-fMRI and combined EEG-MEG-fMRI, the investigators will investigate TC dysconnectivity (fMRI) and alpha dysrhythmia (EEG/MEG) during experimental pressure pain and chronic back pain.

ELIGIBILITY:
Healthy subjects for both MGH and FSU sites

Inclusion Criteria:

1. healthy male and female adults
2. Between the ages of 18 and 60 years
3. Meeting the MRI / MEG / EEG screening criteria
4. Fluent in English; English can be a second language provided that the patients understand all questions used in the assessment measures. This will be asked and judged during the phone screen.

Exclusion Criteria:

1. Current or past history of major medical, neurological, or psychiatric illness based on self-report
2. History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome (for example: asthma or claustrophobia)
3. History of head trauma
4. Pregnant or lactating
5. Presence of any contraindications to MRI scanning (for example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, cannot lie still in fMRI scanner)
6. Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
7. Active substance abuse disorders (based on subject self-report)

Subjects with chronic low back pain (MGH site)

Inclusion Criteria:

1. Volunteers 18-60 years of age
2. Meet the Classification Criteria of the chronic LBP (having low back pain for more than 6 months)
3. At least 4/10 clinical pain on the 0-10 LBP NRS
4. Meeting the MRI / MEG / EEG screening criteria
5. Fluent in English; English can be a second language provided that the patients understand all questions used in the assessment measures. This will be asked and judged during the phone screen.

Exclusion Criteria:

1. Specific causes of back pain (eg, cancer, fractures, spinal stenosis, infections)
2. Complicated back problems (eg, prior back surgery, medicolegal issues)
3. The intent to undergo surgery during the time of involvement in the study
4. Current or past history of major medical, neurological, or psychiatric illness based on self-report
5. History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome (for example: asthma or claustrophobia)
6. History of head trauma
7. Pregnant or lactating
8. Presence of any contraindications to MRI scanning (for example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, cannot lie still in fMRI scanner)
9. Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
10. Active substance abuse disorders (based on subject self-report)
11. Regular use of pain medication such as opioids, nonopioid analgesics, coanalgesics, corticosteroids, or immunomodulatory agents
12. Current use of psychotropic medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects and individuals with chronic low back pain
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
thalamocortical functional connectivity | baseline
  functional connectivity between the thalamus and cortex as measured by resting state fMRI
alpha oscillations | baseline
  alpha oscillations as measured by EEG and MEG

SECONDARY OUTCOMES:
alpha band source | Baseline
  MEG and EEG data will be used to estimate the alpha band source

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Massachusetts General Hospital, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No